CLINICAL TRIAL: NCT03040453
Title: Comparison of Immunological Response After Microwave Ablation and Irreversible Electroporation of Hepatocellular Carcinoma
Brief Title: Immunological Response After Ablative Therapy in the Liver
Acronym: IRAL
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: poor recruitment
Sponsor: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EPN 2016/2212-31/2
Record Dates: First submitted 2017-01-20; First posted 2017-02-02 (Estimated); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Hepatocellular Carcinoma; Immune Response
Keywords: Irreversible electroporation; Microwave ablation
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Electroporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microwave ablation (Other): 20 patients will be treated with microwave ablation
  Interventions: Device: Microwave ablation
- Irreversible electroporation (Other): 20 patients will be treated with irreversible electroporation
  Interventions: Device: Irreversible electroporation

INTERVENTIONS:
Device: Microwave ablation
  Arms: Microwave ablation
Device: Irreversible electroporation
  Other Names: Nano Knife, Angiodynamics
  Arms: Irreversible electroporation

SUMMARY:
Local ablative treatment of Hepatocellular Carcinoma is performed primary on patients not eligible for liver transplant or liver resection. At our Hospital two different methods are used: Microwave ablation, where the tumor cells are heated up and killed, and Irreversible electroporation, where the tumor cells are exposed to an electrical field and nano-pores are formed in the cell membranes and the cells go into apoptosis (programed cell death).

Previous studies have shown effects on the immune system after ablative therapies.

The purpose of this study is to compare the immunological response after the wo different methods of killing the tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular carcinoma, maximum 3 lesions, maximum 30 mm in any cross section diameter
* Physically fit to undergo general anaesthesia
* Fully understand swedish instructions regarding the study

Exclusion Criteria:

* Atrial fibrillation (for irreversible electroporation)
* Pacemaker (for irreversible electroporation)
* >3 lesions
* > 30 mm in any cross section diameter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Immunological response | Change from baseline (morning of the procedure) measured at post operative day 1,7, 28 and 90
  Change in immunological response

SECONDARY OUTCOMES:
Number of participants with complete radiological response at follow up 3, 6, 9 and 12 months. | Follow-up every three months for one year with CT scan.
  Compare the effect of the two different ablative methods

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Freedman, MD, PhD, Principal Investigator — Karolinska Instituet
Locations (1):
- Department of Surgery and Urology, Danderyd Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No